CLINICAL TRIAL: NCT04643704
Title: Evaluation of Quality of Life and Eating Disorders in Children With Food Protein Induced Enterocolitis Syndrom, Food Allergy or Celiac Disease
Brief Title: Quality of Life and Eating Disorders in Children With FPIES, Food Allergy or Celiac Disease
Acronym: QUALIM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201063; IDRCB 2020-A02017-32 (Other: ANSM)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: FPIES; IgE Mediated Food Allergy; Celiac Disease
Keywords: Quality of life; Food avoidance; restriction; Food allergy; Feeding disorder; Psychology
MeSH Terms: conditions — Food Hypersensitivity; Celiac Disease; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- FPIES: 100 patients
- IgE mediated food allergy: 100 patients
- Celiac disease: 100 patients
- Control group: 100 patients

SUMMARY:
Food allergies are associated with a decrease in quality of life. Patients with FPIES often have more food avoidance than necessary. The greater the number of avoided foods, the greater the risk of eating disorders.

To date, no study about quality of life or assessment of eating difficulties has been performed in a French-speaking pediatric population with FPIES or celiac disease

DETAILED DESCRIPTION:
1.1 Current state of knowledge

IgE-mediated food allergies are allergies whose symptoms are urticaria, angioedema, rhinoconjunctivitis, digestive signs, bronchospasm, or even anaphylaxis within 2 hours after ingestion of food. The prevalence of these food allergies in children ranges from 1.6% to 5.6%. Patients with food allergy should follow a strict avoidance diet of the culprit food, until tolerance get acquired in a few months or years later. The avoidance diet is set up by the parents, and must be applied in all places where the child lives (family, nursery and school). Careful reading of the labels and displays in collective restorations are essential in order to limit accidental ingestion. For the most ubiquitous and / or risky foods, parents often have to provide packed lunches. An IgE-mediated emergency kit is required, containing an antihistamine, and sometimes a self-injectable epinephrine pen and bronchodilators. The protocol in the event of an allergic reaction must be known by all caregivers for the child, in order to react immediately if necessary.

Food protein-induced enterocolitis syndrome or FPIES is one of the non IgE-mediated forms of food allergy. Incidence is estimated around 0.015-0.7% in infants and children. FPIES symptoms are delayed: vomiting within 1 to 4 hours after ingestion of the offending food, associated with other symptoms such as lethargy with pallor, diarrhea secondarily. Unlike other non IgE-mediated allergies, FPIES is a potentially severe allergy, with hypovolemic shock seen in 15-33% of cases with dehydration. The most frequently offending foods are ubiquitous, such as milk, fish, eggs, rice and oats. The management of patients with FPIES consists of the avoidance of the offending food(s) until that tolerance is acquired spontaneously in a few months or years. A specific first aid kit is also prescribed, in order to limit dehydration in the event of vomiting after an accident of ingestion, with at least oral rehydration solution.

Celiac disease is a gluten-induced autoimmune enteropathy responsible for digestive malabsorption. It affects 1.4% of the population in the world. The symptoms are very varied, such as chronic diarrhea or chronic constipation resistant to laxative treatment, abdominal distension, chronic fatigue, weight loss and growth retardation, nutritional deficiencies. The treatment consists of a lifelong elimination of gluten only (strict for wheat, rye, barley, and controlled for oats). To date, celiac disease is not curable, but the elimination diet allows clinical, biological and histological normalization in the digestive mucosa. Unlike FPIES or IgE-mediated allergies, the patient and their family do not have to fear a severe reaction in case of accidental exposure, and no first aid kit is required.

1.2 Description of the population to be studied and justification of their choice

FPIES and IgE-mediated food allergies primarily affect young children. A limiting factor in terms of age for this study is the fact that the Food Allergy Quality of Life Questionnaire (FAQLQ) has not been translated into French for adolescents over 12 years old.

The population studied is therefore children under 12 years of age, with a diagnosis of FPIES, IgE-mediated allergy or celiac disease. A control group is also planned to be included.

1.3 Description of the elements covered by the study

. Quality of Life

Food allergies negatively impact the quality of life of patients and their families due to prolonged and restrictive avoidance diet.

The quality of life of children with celiac disease does not differ from that of healthy children.

In our experience, parents of patients with FPIES often report fear of another impressive allergic reaction, with profuse vomiting, and a child described as lethargic and pale during the reaction.

Parents sometimes prefer to delay entering the community in the face of fear of accidental exposure to the culprit allergen, or the fear of a reaction with the introduction of new food, especially if the child is already allergic to several groups of food.

The quality of life of families is more impaired in cases of FPIES than in cases of IgE-mediated food allergy.

During childhood, there are 2 ways to assess the quality of life: a) by measuring the quality of life of the child himself, or b) by measuring the quality of life of the child according to the perception of parents.

The generic PedsQLTM quality of life questionnaire was validated in English and in French to assess children's quality of life, using a form to be completed by parents from birth and / or by the child after the age of 5.

Food allergy-specific quality of life questionnaires: FAQL-PB (Food Allergy Quality of Life-Parental Burden) and FAQLQ-PF (Food Allergy Quality of Life Questionnaire - Parent Form) have been validated for IgE-mediated food allergies and in FPIES in parents of children aged 0 to 12 in an English version. There is also a French version of FAQLQ-PF and FAQLQ-CF (Food Allergy Quality of Life Questionnaire - Child Form).

To date, no quality of life study has been performed in a French-speaking pediatric population with FPIES or celiac disease.

Eating disorders

Food neophobia is physiological between the ages of 2 and 6, but becomes pathologic if it persists beyond 6 years or if it is exacerbated between 2 and 6 years. It is defined by a refusal to eat foods which are new or not known by the child.

Although the majority of patients with FPIES are allergic to only one food, children's diets are often over-restricted to several food groups.

Eating disorders affect 22 to 50% of children with FPIES. These are mainly food refusals, swallowing or chewing difficulties, and sensory disturbance. The risk of food refusal is increased in the event of multiple-food FPIES. In a cohort of 32 patients, only half of these patients received a specialist opinion for the management of eating disorders, probably due to default screening for these disorders.

The French Child Food Rejection Scale (CFRS) score allows screening for food neophobia and pickiness in children aged 2 to 7.

For older children (over 7 years old) and adults, there is the Food Neophobia Scale (FNS), adapted in French (AFNS: Adapted Food Neophobia Scale).

To date, no study has evaluated eating disorders in a French-speaking pediatric population with FPIES or celiac disease.

1.4 Rationale for the duration of the study The research will last at least 2 years. The goal is to include at least 100 patients with FPIES, 100 patients with IgE-mediated food allergy other than FPIES, 100 patients with celiac disease and 100 control patients.

ELIGIBILITY:
Inclusion Criteria:

Any patient from 0 to 12 years of age, with FPIES or an IgE-mediated food allergy or celiac disease.

Controls: chid from 0 to 12 years old, without any food avoidance for medical reason, and without chronical severe pathology

Exclusion Criteria:

General exclusion criteria:

* Families and patients who do not understand French
* Cured food allergy (FPIES, IgE or non IgE-mediated food allergy)
* Allergic patient (FPIES, IgE-mediated food allergy) undergoing oral or epicutaneous tolerance induction

Criteria for non-inclusion in the "FPIES" group:

* Patient with mixed FPIES with associated IgE-mediated symptomatology
* Non IgE-mediated food allergies other than FPIES

Criteria for non-inclusion in the "celiac disease" group:

- Patient with hypersensitivity to non-celiac gluten

Criteria for non-inclusion in the "control" group:

* Current food avoidance, personal or in one of the household members due to allergy, or digestive disorders (abdominal pain, diarrhea for example) induced by the consumption of particular foods and requiring a strict avoidance diet
* Chronic digestive pathology (chronic inflammatory bowel disease, functional bowel disorders with a correlation of symptoms with diet, esophagitis and eosinophilic enteropathy)
* Chronic nutritional, metabolic or endocrine pathologies for which diet can have an impact: obesity, dyslipidemia, diabetes
* Severe chronic respiratory pathology (eg: cystic fibrosis, chronic respiratory failure)

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients recruited from hospitalization (conventional, and day-care unit) and consultation.
  Healthy controls without any food avoidance recruited from consultations, hospitalisations or community.
  Multicentric study
  * Pediatric Nutrition and Gastroenterology Unit - Trousseau Hospital, APHP;
  * Pediatric Pneumology and Allergy Unit - Necker-Enfants Malades Hospital, APHP;
  * Pediatric department and Asthma and Allergy unit - Ambroise Paré Hospital, APHP.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) in children with FPIES | 12 months
  FAQLQ (Food Allergy Quality of Life Questionnaire)-PF (Parent form) for parents of children from 0 to 12 years old with FPIES FAQLQ-CF (Child Form) for children between 8 to 12 years old with FPIES PedsQLTM: generic questionnaire of QoL for parents and children from 0 to 12 years old with FPIES

SECONDARY OUTCOMES:
Food neophobia in children with FPIES | 24 months
  CFRS (Child Food Rejection Scale) for children with FPIES from 2 to 7 years old AFNS (Adapted Food Neophobia Scale) for children with FPIES from 8 to 12 years old
QoL in children with food allergy | 24 months
  FAQLQ-PF for parents of children from 0 to 12 years old with IgE-mediated food allergy FAQLQ-CF for children between 8 to 12 years old with IgE-mediated food allergy PedsQLTM: generic questionnaire of QoL for parents and children from 0 to 12 years old with IgE-mediated food allergy
QoL in children with celiac disease | 24 months
  : generic questionnaire of QoL for parents and children from 0 to 12 years old with IgE-mediated food allergy PedsQLTM child form: generic questionnaire of QoL for children from 5 to 12 years old
QoL in children without any food avoidance | 24 months
  PedsQLTM: generic questionnaire of QoL for parents and children from 0 to 12 years old with IgE-mediated food allergy PedsQLTM child form: generic questionnaire of QoL for children from 5 to 12 years old
Food neophobia in children with food allergy | 24 months
  CFRS (Child Food Rejection Scale) for children from 2 to 7 years old AFNS (Adapted Food Neophobia Scale) for children from 8 to 12 years old
Food neophobia in children with celiac disease | 24 months
  CFRS (Child Food Rejection Scale) for children from 2 to 7 years old AFNS (Adapted Food Neophobia Scale) for children from 8 to 12 years old
Food neophobia in children without any food avoidance | 24 months
  CFRS (Child Food Rejection Scale) for children from 2 to 7 years old AFNS (Adapted Food Neophobia Scale) for children from 8 to 12 years old

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Lemoine, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Trousseau Hospital, Service : Nutrition et Gastroentérologie Pédiatrique, Paris, France

IPD SHARING:
Plan to Share IPD: Yes